CLINICAL TRIAL: NCT03722680
Title: Effectiveness Assessment of Riluzole in the Prevention of Oxaliplatin-induced Peripheral Neuropathy: A Phase II Randomized Study by UNICANCER With the Cooperation of AFSOS
Brief Title: Effectiveness Assessment of Riluzole in the Prevention of Oxaliplatin-induced Peripheral Neuropathy.
Acronym: RILUZOX-01
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of treatment, sponsor decision.
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UC-0106/1712; 2017-002320-25 (EudraCT Number)
Record Dates: First submitted 2018-10-11; First posted 2018-10-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-10

CONDITIONS: Oxaliplatin-induced Peripheral Neuropathy
Keywords: Riluzole; oxaliplatin; colorectal cancer; neuropathy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: Riluzole arm: The patient will be taken one tablet (riluzole 50 mg, film-coated tablet) twice a day, in the morning and in the evening during the meal (12h interval). The medication is taken during the 14 days of each chemotherapy cycle, beginning 7 days before the start of chemotherapy and ending 2 weeks after the start of last cycle of chemotherapy (25 weeks). The treatment ends with the cessation of chemotherapy (visit V3 or anticipated stop).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo arm: The patient will be taken on tablet (placebo :50 mg, film-coated tablet) Posology, administration and duration of treatment will be equivalent to riluzole group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riluzole (Experimental): The patient will be taken one tablet twice a day, in the morning and in the evening during the meal (12h interval). The medication is taken during the 14 days of each chemotherapy cycle, beginning 7 days before the start of chemotherapy and ending 2 weeks after the start of last cycle of chemotherapy (25 weeks). The treatment ends with the cessation of chemotherapy (visit V3 or anticipated stop).
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator): Posology, administration and duration of treatment will be equivalent to riluzole group.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Riluzole — Riluzole during chemotherapy (oxaliplatin)
  Arms: Riluzole
Drug: Placebo Oral Tablet — placebo
  Arms: Placebo

SUMMARY:
It is a phase II trial, randomized, parallel, double blind, multicenter, comparing riluzole versus placebo.

The trial population is composed of patients ≥18 years old that have developed stage II/III colorectal cancer and are eligible for Simplified FOLFOX4 (6-12 cycles) adjuvant chemotherapy.

The primary objective is to assess the preventive efficacy of riluzole on the severity of oxaliplatin-induced peripheral neuropathy during the Simplified FOLFOX4 adjuvant chemotherapy of stage II/III colorectal cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years old,
2. Eligible patient starting adjuvant oxaliplatin-based chemotherapy (6-12 cycles, Simplified FOLFOX4) for stage II/III colorectal cancer,
3. Histological or cytological confirmation of colorectal cancer,
4. Performance status (ECOG) ≤2,
5. Normal hematological function (ANC ≥1.5 x 10⁹/L; platelets count ≥100 x 10⁹/L; hemoglobin ≥9.0 g/dL),
6. Normal hepatic function: total bilirubin ≤1.5 x upper limit of normal (ULN) (unless documented Gilbert's syndrome); aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤3 x ULN, and gamma-glutamyltransferase (GGT) ≤3 x ULN,
7. Normal renal function: serum creatinine ≤1.5 x ULN,
8. Normal cardiac function: ECG,
9. Patients affiliated to the French national health insurance,
10. Patient must have signed a written informed consent form prior to any study specific procedures,
11. French language comprehension,
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Metastatic cancer,
2. Diagnosis of neuropathy,
3. EORTC QLQ-CIPN20 sensory score >6,
4. Previous neurotoxic chemotherapy treatment,
5. Patients with chronic obstructive pulmonary disease,
6. ALAT/ASAT elevated more than 3 times the normal value,
7. Patients with known allergy or severe hypersensitivity to riluzole or any of the study drug excipients,
8. Dependence on alcohol or drugs,
9. Psychotic disorders,
10. Women pregnant or breastfeeding,
11. Patients undergoing a measure of legal protection (trusteeship, guardianship ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire-chemotherapy-induced peripheral neuropathy (QLQ-CIPN20) | 3 months afer initiation of oxaliplatin based chemotherapy (1 cycle = 14 days)
  QLQ-CIPN20 Questionnaire (EORTC):
  Self-reported questionnaire consisting of 20 questions that assess the symptoms and functional limitations of chemotherapy-induced peripheral neuropathy. The questionnaire is divided in 3 subscales: sensory, motor, and autonomic and gives a comprehensive picture of the nature, frequency, and severity of chemotherapy-induced peripheral neuropathy (CIPN). Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), patients indicate the degree to which they have experienced sensory, motor, and autonomic symptoms.

SECONDARY OUTCOMES:
QLQ-CIPN20 | At inclusion (V0), 3 months (V2), up to 7 months (V3), up to 9 months (V4), up to 12 months (V5), up to 15 months (V6), and up to 18 months (V7) after initiation of oxaliplatin based chemotherapy.
  Self-reported questionnaire consisting of 20 questions that assess the symptoms and functional limitations of chemotherapy-induced peripheral neuropathy. The questionnaire is divided in 3 subscales: sensory, motor, and autonomic and gives a comprehensive picture of the nature, frequency, and severity of CIPN. Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), patients indicate the degree to which they have experienced sensory, motor, and autonomic symptoms.
National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | throughout study completion, assessed up to 43 months
  The NCI-CTCAE v5.0 is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale will assess the severity of sensory neuropathic disorders, this derivative into 5 grades determined by the investigator.
Brief Pain Inventory (BPI) questionnaire | At inclusion (V0), 3 months (V2), up to 7 months (V3), up to 9 months (V4), up to 12 months (V5), up to 15 months (V6), and up to 18 months (V7) after initiation of oxaliplatin based chemotherapy.
  This self-report questionnaire includes:
  * A body schema
  * The maximum pain, lowest pain, usual pain within the last 15 days (Numerical Numeric rating scales (NRS) 0 to 10
  * Description of current analgesic treatment,
  * An assessment of relief by a percentage scale (0-100%), Assessment of the impact of pain on: mood, relationships with others, walking, sleep, work, happiness the joy - of living, recreation, activities in general (digital scales, rating from 0 [normal] to 10 [no activity]).
Douleur Neuropathique 4 (DN4) questionnaire (interview portion) | This evaluation will be carried out only if the item 5 of BPI "general pain felt in the last 7 days" is ≥4/10.
  The interview portion of the DN4 questionnaire is a clinician-administered screening tool for neuropathic pain. The questionnaire includes 7 items, grouped into two questions. Each item, is answered as either YES or NO. A final cumulative patient's score is obtained by allocating 1 point for each YES and 0 point for each NO. If the patient's score is ≥3/7, the test is positive.
Neuropathic Pain Symptom Inventory (NPSI) questionnaire | This evaluation will be carried out only if the item 5 of BPI "general pain felt in the last 7 days" is ≥4/10.
  This self-reported questionnaire assesses different neuropathic pain symptoms. The French NPSI includes 12 items that discriminates and quantifies five distinct dimensions of neuropathic pain. Each of these items are quantified on a (0-10) numerical scale.
QLQ-C30 questionnaire (EORTC) | At inclusion (V0), 3 months (V2), up to 7 months (V3), up to 9 months (V4), up to 12 months (V5), up to 15 months (V6), and up to 18 months (V7) after initiation of oxaliplatin based chemotherapy.
  This self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Disease progression | From date of randomisation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 43 months.
  Disease Free Survival, defined as the interval between the date of randomization and the date of cancer relapse (local, regional, metastases, second cancer) or death from any cause, whichever occurs first.
Time to HRQoL score deterioration | At inclusion (V0), 3 months (V2), up to 7 months (V3), up to 9 months (V4), up to 12 months (V5), up to 15 months (V6), and up to 18 months (V7) after initiation of oxaliplatin based chemotherapy.
  The interval between randomization and deterioration ≥5 points in the HRQoL score as compared to baseline score or death (all causes).
Quantification of chemotherapy dose reductions | 3 months (V2) and up to 7 months (V3) after initiation of oxaliplatin based chemotherapy.
  The number of chemotherapy dose reduction caused by severe neuropathy and/or poor tolerance of treatment will be recorded.
Quantification of cumulative dose | 3 months (V2) and up to 7 months (V3) after initiation of oxaliplatin based chemotherapy.
  The cumulative dose (mg/m²) of chemotherapy delivered to patients will be recorded.
Evaluation of study exit rates | 3 months (V2) and up to 7 months (V3) after initiation of oxaliplatin based chemotherapy.
  The study exit rate caused by severe neuropathy and/or poor tolerance of treatment will be recorded.
Assessment of glutamate serum level | Glutamate serum level will be dose at inclusion (V0), 3 months (V2), up to 7 months (V3), and up to 18 months (V7) after initiation of oxaliplatin based chemotherapy.
  Correlation with colorectal cancer tumors/nodes/metastases (TNM) score (and eventually neuropathic symptoms), glutamate plasmatic

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - ICO - Site Paul Papin, Angers
  - CH Beauvais, Beauvais
  - Centre François Baclesse, Caen
  - Hia Percy, Clamart
  - CHU de Clermont -Ferrand, Clermont-Ferrand
  - Clinique St Côme, Compiègne
  - GHPSO, Creil
  - Centre Georges François Leclerc, Dijon
  - CHU de Dijon, Dijon
  - CH Annecy-Genevois, Pringy
  - CHU de Reims, Reims
  - Institut Jean Godinot, Reims
  - ICO - Site René Gauducheau, Saint-Herblain
  - Hia Begin, Saint-Mandé
  - CHU de Saint-Etienne, Saint-Priest
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Kerckhove N, Busserolles J, Stanbury T, Pereira B, Plence V, Bonnetain F, Krakowski I, Eschalier A, Pezet D, Balayssac D. Effectiveness assessment of riluzole in the prevention of oxaliplatin-induced peripheral neuropathy: RILUZOX-01: protocol of a randomised, parallel, controlled, double-blind and multicentre study by the UNICANCER-AFSOS Supportive Care intergroup. BMJ Open. 2019 Jun 9;9(6):e027770. doi: 10.1136/bmjopen-2018-027770. PMID 31182448